CLINICAL TRIAL: NCT00834821
Title: Integrated Multi-setting Psychosocial Treatment for ADHD-Inattentive Type
Brief Title: Effectiveness of a Behavioral Treatment Program for Attention Deficit Hyperactivity Disorder, Inattentive Type
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R01MH077671 (NIH); R01MH077671 (NIH); DSIR 84-CTS
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Hyperactivity Disorder; ADHD, Predominantly Inattentive Type; Inattention; Psychosocial Intervention; Behavioral Intervention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Participants will undergo the Child Life and Attention Skills (CLAS) Program.
  Interventions: Behavioral: Child Life and Attention Skills (CLAS) Program
- 2 (Active Comparator): Participants will undergo parent focused training (PFT).
  Interventions: Behavioral: Parent Focused Training (PFT)
- 3 (No Intervention): Participants will receive a list of referrals for clinical services as needed, including professional organizations, support groups, and the community mental health system.

INTERVENTIONS:
Behavioral: Parent Focused Training (PFT) — PFT will involve parenting skills training supplemented with a phone session between a therapist and teacher to cover ADHD, inattentive type. This intervention will include ten 90-minute parent group training sessions and up to five individual sessions with the study therapist.
  Arms: 2
Behavioral: Child Life and Attention Skills (CLAS) Program — CLAS will involve parenting skills training adapted for ADHD, inattentive type; child life skills training; and teacher consultation. This intervention will include ten 90-minute parent group training sessions; ten 90-minute child group training sessions; up to five individual family sessions with the study therapist; and up to six 30-minute sessions with the teacher, parent, and therapist.
  Arms: 1

SUMMARY:
This study will test the effectiveness of a new behavioral treatment, called the Child Life and Attention Skills Program, for children with attention deficit hyperactivity disorder, inattentive type.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is a common childhood disorder in which problems with focusing disrupt a normal life. There are two subtypes of ADHD: combined type (ADHD-C), which includes symptoms of inattention and hyperactivity or impulsivity, and inattentive type (ADHD-I), in which symptoms are limited to inattention. The profile of ADHD-I, including attention deficits, comorbid disorders, social impairments, and neurocognitive functioning, is sufficiently different from the profile of ADHD-C that treatments effective for ADHD-C may not also be effective in treating ADHD-I. Most studies of ADHD treatment evaluate ADHD-C, and there is very little research into treatments aimed specifically at ADHD-I. The Child Life and Attention Skills (CLAS) Program is a behavioral program designed specifically for ADHD-I and combines life skills training for the child, teacher consultation, and parent training techniques adapted from ADHD-C treatments. This study will compare the effectiveness of the CLAS Program, standard parent training, and community referrals in treating children with ADHD-I.

Participation in this study will last 11 to 12 weeks, followed by a 5- to 7-month follow-up period. On the basis of parent and teacher evaluations of each child's behavior, invitations to participate in screening procedures for the study will be extended to children and their parents. There will be two screening visits, during which the child will undergo reviews of medical and developmental history, diagnostic interviews, intelligence testing, academic achievement testing, and neuropsychological testing. The child and parent will be videotaped in a series of interactions, and both will complete questionnaires about child functioning, parent functioning, family functioning, and family relations. The child's teacher and school principal will also be contacted to ensure that they are willing to participate in the study.

Eligible participants will then be randomly assigned to receive the CLAS Program, parent-focused training (PFT), or community referrals. The CLAS Program will involve a half-hour orientation and up to five half-hour weekly meetings with the child's teacher, therapist, and parent over 11 to 12 weeks. The program will also involve ten 1.5-hour group sessions for parents, with separate group sessions for children at the same time, and up to five individual family sessions led by a therapist. Teachers will participate in a school-home note system for maintaining and rewarding child behavior; parents will be taught strategies for giving commands, using rewards and consequences, and establishing routines and organizational schemes; and children will be taught social interaction skills, homework skills, and organizational skills.

Participants in the PFT group will attend the ten 1.5-hour parent group sessions and up to five individual family sessions. Participants in the community referrals group will only receive referrals to community mental health practitioners.

All participants will undergo assessments that are similar to those in the screening visit after completing treatment and again at a follow-up visit 5 to 7 months later. Participants in the CLAS and PFT groups will continue monthly individual family sessions with a therapist until undergoing the follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Primary DSM-IV diagnosis of attention deficit hyperactivity disorder, inattentive type (ADHD-I)
* IQ score greater than 80
* Living with one biological or adoptive parent for the past year
* Currently attending school full time
* Consent of school to participate in the study

Exclusion Criteria:

* Current use of nonstimulant psychoactive medication
* Severe visual or hearing impairment
* Severe language delay
* Major neurological illness
* Diagnosis of one of the following: psychosis, bipolar disorder, obsessive-compulsive disorder, pervasive developmental disorder, clinical depression, or suicidality
* Enrolled in all-day special education
* Parent or child does not speak English
* Child or family is currently involved in and expects to continue psychotherapy to address child's attention, behavioral, or emotional problems

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 199 (Actual)
Dates: Start 2008-11-01 (Actual); Primary Completion 2013-01-03 (Actual); Study Completion 2013-01-03 (Actual)

PRIMARY OUTCOMES:
Inattention symptoms, as defined by the DSM-IV | Measured immediately post-treatment and at a follow-up 5 to 7 months later

SECONDARY OUTCOMES:
Academic and social functioning | Measured immediately post-treatment and at a follow-up 5 to 7 months later

CONTACTS AND LOCATIONS:
Overall Officials: Linda J. Pfiffner, PhD, Principal Investigator — University of California, San Francisco; Keith McBurnett, PhD, Principal Investigator — University of California, San Francisco; Stephen P. Hinshaw, PhD, Principal Investigator — University of California, Berkeley
Locations (2):
- United States (2):
  - University of California, Berkeley, Berkeley, California
  - University of California, San Francisco, San Francisco, California